CLINICAL TRIAL: NCT01154634
Title: A Double-blind, Randomized, Placebo-controlled, Two-centre, Phase IIa Pharmacodynamic Cross-over Study to Assess the Effect of AZD2516 on the Total Number of Reflux Episodes in Healthy Male Volunteers
Brief Title: Study to Investigate the Pharmacodynamic Effect of a Single Dose of AZD2516 in Healthy Male Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3830C00001
Record Dates: First submitted 2010-06-15; First posted 2010-07-01 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Reflux
Keywords: Pharmacodynamic effect; Reflux inhibition
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- First 5 mg, then placebo, then 16 mg, then 40 mg (Experimental): period 1: AZD2516 5 mg, period 2: washout, period 3: placebo, period 4: washout, period 5: AZD2516 16 mg, period 6: washout, period 7: AZD2516 40 mg.
  Interventions: Drug: AZD2516, 5 mg; Drug: AZD2516, 16 mg; Drug: AZD2516, 40 mg; Drug: Placebo
- First 40 mg, then 16 mg, then placebo, then 5 mg (Experimental): period 1: AZD2516 40 mg, period 2: washout, period 3: AZD2516 16 mg, period 4: washout, period 5: placebo, period 6: washout, period 7: AZD2516 5 mg.
  Interventions: Drug: AZD2516, 5 mg; Drug: AZD2516, 16 mg; Drug: AZD2516, 40 mg; Drug: Placebo
- First 16 mg, then 5 mg, then 40 mg, then placebo (Experimental): period 1: AZD2516 16 mg, period 2: washout, period 3: AZD2516 5 mg, period 4: washout, period 5: AZD2516 40 mg, period 6: washout, period 7: placebo.
  Interventions: Drug: AZD2516, 5 mg; Drug: AZD2516, 16 mg; Drug: AZD2516, 40 mg; Drug: Placebo
- First placebo, then 40 mg, then 5 mg, then 16 mg (Experimental): period 1: placebo, period 2: washout, period 3: AZD2516 40 mg, period 4: washout, period 5: AZD2516 5 mg, period 6: washout, period 7: AZD2516 16 mg
  Interventions: Drug: AZD2516, 5 mg; Drug: AZD2516, 16 mg; Drug: AZD2516, 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: AZD2516, 5 mg — Capsule, oral
Drug: AZD2516, 16 mg — Capsule, oral
Drug: AZD2516, 40 mg — Capsule, oral
Drug: Placebo — Capsule, oral

SUMMARY:
The purpose of this study is to investigate the pharmacodynamic effect of AZD2516 in healthy male subjects.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, two-centre, phase IIa pharmacodynamic cross-over study to assess the effect of AZD2516 on the total number of reflux episodes in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Healthy male subjects
* Age 18-45 years, inclusive

Exclusion Criteria:

* Clinically significant illness within the 2 weeks prior to the first dose of study drug
* History of clinically significant cardiovascular, respiratory, renal, hepatic, neurological, mental or gastrointestinal disease
* Need for concomitant medications during the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berner Hansen, Study Director — AstraZeneca R&D Molndal
Locations (2):
- Research Site, Leuven, Belgium
- Research Site, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 25 participants were enrolled into the study at 2 medical centres (14 and 11 participants), 20 of them were randomised to treatment (10 at each medical centre) and all these 20 participants completed the study.
Pre-assignment Details: After enrolment, participant's eligibility for assignment to treatment was based on inclusion and exclusion criteria.
Period: Period 1 - First Intervention
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 - Washout
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 3- Second Intervention
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 - Washout
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 5 - Third Intervention
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 6 - Washout
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 7 - Fourth Intervention
Arm/Group | First 5 mg, Then Placebo, Then 16 mg, Then 40 mg | First 40 mg, Then 16 mg, Then Placebo, Then 5 mg | First 16 mg, Then 5 mg, Then 40 mg, Then Placebo | First Placebo, Then 40 mg, Then 5 mg, Then 16 mg
Started | 4 | 7 | 4 | 5
Completed | 4 | 7 | 4 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AZD2516 5 mg: Loading dose: 3 * AZD2516 1 mg capsules. Maintenance doses: 1 * AZD2516 1 mg capsule, 2 * placebo capsules and 1 * AZD2516 1 mg capsule, 2 * placebo capsules.
- AZD2516 16 mg: Loading dose: 2 * AZD2516 5mg capsule, 1 * placebo capsule. Maintenance dose: 3 * AZD2516 1 mg capsule and 3 * AZD2516 1 mg capsule.
- AZD2516 40 mg: Loading dose: 2 * AZD2616 10 mg capsules, 1 * placebo capsule. Maintenance dose: 2 * AZD2616 5 mg capsules, 1 * placebo capsule and 2 * AZD2616 5 mg capsules, 1 * placebo capsule.
- Placebo: Loading dose: 3 * placebo capsules. Maintenance dose: 3 * placebo capsules and 3 * placebo capsules.
- Total: Total of all reporting groups
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo | Total
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 20
Age Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 31 (9.6) | 25 (4.5) | 28.8 (5.9) | 23 (4.2) | 26.95 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 7 | 4 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Reflux Episodes 0 to 3 Hours Post Meal
Description: Total number of reflux episodes 0 to 3 hours post meal
Time Frame: 0 to 3 hours post meal
Population: Data from two subjects (one in arm AZD2516 5 mg, and one in arm Placebo) were excluded from efficacy analysis due to incorrect medication received.
Measure: Geometric Mean (Full Range); unit: Episodes
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 19
Episodes | 15.1 [1 to 149] | 12.5 [0 to 50] | 11.0 [0 to 41] | 12.7 [0 to 40]

2. Secondary Outcome: Transient Lower Esophagus Sphincter Relaxations (TLESRs) 0 to 3 Hours Post Meal
Description: Number of TLESRs 0 to 3 hours post meal were calculated based upon the manometric analysis fpr the 3-hour post-meal period.
Time Frame: 0 to 3 hours post meal
Population: Data from two subjects were excluded from efficacy analysis due to incorrect medication received Data from five visits from two subject were excluded form analysis due to deviations caused by technical problems.
Measure: Geometric Mean (Full Range); unit: relaxations
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 18 | 19 | 18 | 18
relaxations | 16.9 [8 to 51] | 16.2 [9 to 26] | 10.4 [2 to 31] | 16.8 [9 to 33]

3. Secondary Outcome: Area Under the Plasma Concentration Curve(AUC)
Description: Area under the plasma concentration vs. time curve from time zero to 12-hours post dose calculated by loglinear trapezoidal method
Time Frame: 0 to 12 hours post dose
Population: Data from one subject in arm AZD2516 5 mg were excluded from efficacy analysis due to incorrect medication received.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol*h/L
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 0
nmol*h/L | 251.5 [188.4 to 335.7] | 906.6 [732.7 to 1122] | 2825 [2185 to 3653] |

4. Secondary Outcome: Average Plasma Concentration (C Average)
Description: Average plasma concentration
Time Frame: 1 to 4 hours post dose
Population: Data from one subject in arm AZD2516 5 mg were excluded from efficacy analysis due to incorrect medication received.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 0
nmol/L | 45.46 [35.04 to 58.98] | 175.8 [142.4 to 217.1] | 506.8 [405.0 to 634.3] |

5. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration
Time Frame: 0 to 12 hours post dose
Population: Data from one subject in arm AZD2516 5 mg were excluded from efficacy analysis due to incorrect medication received.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 0
nmol/L | 103.8 [76.09 to 141.5] | 378.0 [315.0 to 453.5] | 911.7 [767.3 to 1083] |

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration (Tmax)
Time Frame: 0 to 12 hours post dose
Population: Data from one subject in arm AZD2516 5 mg were excluded from efficacy analysis due to incorrect medication received.
Measure: Median (Full Range); unit: hours
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 0
hours | 0.750 [0.500 to 4.000] | 0.750 [0.500 to 1.250] | 1.000 [0.500 to 4.000] |

7. Secondary Outcome: Terminal Half-life (T Half)
Description: Terminal half-life (T half)
Time Frame: 0 to 12 hours post dose
Population: Data from one subject in arm AZD2516 5 mg were excluded from efficacy analysis due to incorrect medication received.
  Two samples were not analyzed for T half due to technical reasons.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 17 | 20 | 20 | 0
hours | 1.221 [1.042 to 1.430] | 1.416 [1.222 to 1.640] | 1.584 [1.414 to 1.774] |

8. Secondary Outcome: Clinically Relevant Change of Laboratory Variables
Description: Number of participants with clinically relevant change of laboratory variables as judged by the responsible medical officer.
Time Frame: Pre-entry to follow-up
Measure: Number; unit: Participants
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | AZD2516 5 mg | AZD2516 16 mg | AZD2516 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 8/20 | 12/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2516 5 mg (N=20) | AZD2516 16 mg (N=20) | AZD2516 40 mg (N=20) | Placebo (N=20)
Disturbance In Attention (Nervous system disorders) | 2 | 5 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 7 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Euphoric Mood (Psychiatric disorders) | 0 | 2 | 2 | 0
Daydreaming (Psychiatric disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days